CLINICAL TRIAL: NCT01299662
Title: An Open Label Study to Evaluate Innate Immune Responses Induced by a Pattern Recognition Receptor Agonist, Poly-ICLC (Hiltonol), in Healthy Volunteers
Brief Title: Polyinosinic-Polycytidylic Acid-poly-L-lysine Carboxymethylcellulose (Poly-ICLC) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MAC-0718
Record Dates: First submitted 2011-02-14; First posted 2011-02-18 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Poly ICLC (Experimental): One 1.6 mg subcutaneous injection of the adjuvant, poly ICLC, in the upper arm.
  Interventions: Drug: Poly ICLC

INTERVENTIONS:
Drug: Poly ICLC — One 1.6 mg subcutaneous injection of the study drug, poly ICLC in the upper arm.

SUMMARY:
Vaccines induce protective immunity against numerous infectious diseases. However, current vaccines have limited efficacy against challenging infections like tuberculosis, malaria, and HIV. Protein vaccines are safe but, typically they induce weak T cell immunity when administered alone. Therefore, special attention is being given to adjuvants, which are enhancers of immunity, that cab mature antigen presenting immunostimulatory dendritic cells. Our goal is to study in humans the mechanism whereby a synthetic adjuvant, poly ICLC, which acts on defined pattern recognition receptors, enhances T an B cell immunity. In preclinical studies, our lab has found in mice that poly IC and its analog poly ICLC are superior adjuvants for T cell mediated immunity relative to other agonists for PRR. Poly ICLC has been extensively studied in humans with a favorable safety profile. In a recently completed Phase I study, poly ICLC was found to be safe and well tolerated when administered as a single dose of 1.6 mg subcutaneously and intranasally to healthy volunteers. In additional, preliminary data shows marked upregulation of gene expression in whole PBMSc following s.c. injection of poly ICLC as well as activation of various blood cell type, including dendritic cells and monocytes. In this study the investigators propose to extend the evaluation of innate immune responses following s.d. injection of poly ICLC to healthy volunteers. The investigators propose to characterize poly ICLC effects on specific blood cell types, focusing on three different subsets of DC's, by analyzing gene transcriptional changes at baseline and at one day following its administration. In order to study the early local effects of poly ICLC, which are important for the recruitment and activation of antigen presenting cells, the investigators also propose to perform skin biopsies at a skin site contralateral to the injection site and at the injection site after poly ICLC injections.

DETAILED DESCRIPTION:
This protocol will take a systems biology approach to understand in humans a major new area of vaccine biology: the mechanism whereby adjuvants, acting on defined pattern recognition receptors [PRR], enhance T and B cell immunity. Our focus is on synthetic double stranded RNA, or poly IC and its more RNase resistant form, called poly ICLC, which is available for studies in humans. The PRRs are the cytosolic helicase, MDA-5, and the endosomal toll like receptor, TLR3. The Steinman lab has pioneered in mice and monkeys that dsRNA is a superior adjuvant for T cell mediated immunity relative to several PRR agonists (Longhi et al., 2009; Stahl-Hennig et al., 2009). A major mechanism is that poly IC is a superior inducer of systemic type I interferon [IFN], which in turn acts on type I IFN receptors [IFNAR] to mature immune stimulatory function of dendritic cells [DCs]. An adaptive Th1 type T cell response is induced, but it is independent of IL-12 and IFN-g.

Multiparameter approaches now provide the means to understand adjuvant action. We hypothesize that DCs undergo changes that are adjuvant-specific and then link innate to select forms of adaptive immunity. Transcriptional arrays of splenic DCs in mice show that dsRNA induces a massive response with ~1000 splenic DC genes changing >2 fold in 4 hrs. These changes are driven primarily via type I IFN, produced systemically via MDA-5 in non-bone marrow derived cells and then acting on DC IFNAR. IFNAR mediate most changes termed "DC maturation" and acquisition of immune stimulating activity, e.g., high CD86, CD40, IL-15, and mechanisms to restore homeostasis. In other words, IFN rather than PRR per se, accounts for the bulk of the poly IC response in DCs.

In a recently completed phase I study (protocol MAC-682), poly ICLC was found to be safe and well tolerated when administered as a single dose of 1.6 mg subcutaneously (s.c.) and intranasally (i.n.) to healthy volunteers. Preliminary innate immune response data shows, similarly to preclinical studies in mice, marked upregulation of gene expression in whole PBMCs following s.c injection of poly ICLC. At day 1 following poly ICLC injection, over 2,000 genes are upregulated (> 1.3 fold change of expression at day 1 versus at baseline) and these responses are specific to the study drug. Importantly, gene changes are homogenous among the 8 volunteers who received poly ICLC. The top upregulated genes are interferon-stimulated genes as it would be predicted since poly ICLC is known to induce type I interferons. In addition, genes associated with dendritric cell (DC) activation such as CD40 and CD86 are also upregulated at day 1 after poly ICLC injection, as well as genes involved in signaling pathways such as IRF 5, IRF 7 and STAT1. Poly ICLC induced secretion of small amounts of types I and II interferons in plasma and these levels peaked at day 2 post injection. Lastly, FACS analysis of PBMCs demonstrated that poly ICLC induced upregulation of activation markers on different subsets of blood dendritic cells. Evaluation of later timepoints are currently taking place but analyses of samples from day 7 show that genes involved in the generation of T and B cell responses are upregulated and the early interferon-stimulated genes are trending down to baseline levels of expression. These results so far show that subcutaneous injection of poly ICLC led to systemic innate immune responses, dominated by the induction of type I interferons. Assays have been performed in whole PBMCs however genetic expression patterns of different subsets of blood leukocytes in response to poly ICLC remain to be defined. We now propose to extend the analysis of systemic immune responses after poly ICLC to the characterization of its transcriptional effects on specific FACS sorted blood cell types, such as DCs, monocytes, NK cells as well as T and B cells. By analyzing individual cell subsets we expect to better dissect how poly ICLC modulates innate immune responses that can in turn affect adaptive immune responses when given in combination with an antigen.

Significant regulation of interferon genes (both type I IFNs and IFN-gamma) was not evident by gene array analysis of whole PBMC's, despite measurement of small amounts of both IFN-alpha and IFN-gamma in plasma. It may be that the platform used was not sensitive enough to detect regulation of IFN genes and we plan to perform RT-PCR to verify these findings. However, it may be that when we restrict our analysis to peripheral blood, we miss the early events that take place following poly ICLC administration. In order to understand how poly ICLC activates different cell populations, it is important to characterize its immunoregulatory effects both locally and systemically.

The cutaneous immune environment is particularly amenable to PRR ligand modulation as evidenced by imiquimod, which acts on TLR 7. Indeed, use of imiquimod to stimulate immune responses against both infectious agents (HPV) and malignancy (squamous and basal cell carcinoma) has been documented. Migratory DCs, which traffic from the skin to the skin draining LN, have been shown to cross prime immune reponses to self and viral antigens. As such, it is possible that skin DCs may migrate into skin draining LNs or blood following poly ICLC administration. However analysis of blood populations alone will likely miss the window of immune alteration if these events are occuring locally in the skin. Analysis of genetic expression and of cellular infiltrates at the site of poly ICLC injection, both early on (at 6 hours) and when skin infiltration is evident clinically (at day 1), will likely add to our understanding of its adjuvant effects. Genomic expression profiles of skin samples have been successfully used for disease classification and to predict response to treatment in skin diseases such as psoriasis and squamous cell carcinoma (Zaba L et al., 2007; Suarez-Farinas et al., 2010). Analysis of genomic expression profile in skin after poly ICLC may prove useful to understand how innate immune responses are initiated by PRRs ligands and perhaps by other vaccine adjuvants.

Most studies of poly ICLC in humans used the intramuscular route of administration. Subcutaneous administration of poly ICLC has not been studied extensively and protocol MAC-682 was the first study to use this route of administration in healthy volunteers. Following poly ICLC s.c. injection, 8 out of 8 volunteers developed a well-defined area of erythema, with some degree of induration and tenderness. This injection site reaction usually peaks at day 2 and is completely resolved by day 7. Histologic data characterizing this infiltrate is not available in humans. However, data is available in non-human primates.

A GLP-compliant toxicology study was performed in cynomolgus macaques to investigate the safety of anti-DEC-205 (3G9) - HIV gag p24 (DCVax-001) in combination with the adjuvant Hiltonol (poly ICLC) subcutaneously. In this study, macaques were administered a total of four doses of 10 mg of anti-DEC-205-HIV gag p24 antibody in combination with 2 mg of poly ICLC, 10 mg of poly ICLC alone or placebo, over 8 weeks. With regard to reactogenicity (modified Draize scoring), there was evidence to indicate that poly ICLC (10 mg) induced very slight and transient injection site reaction in the form of erythema; however, the reaction was reduced or absent with repeated dosing, indicating that it was of minimal toxicological significance. A number of gross lesions including dark area, dark discoloration or gelatinous material were present in the most recent site of administration prior to euthanasia, 1 day after poly ICLC injection. At least one of these findings occurred in all animals of both genders receiving 10 mg poly-ICLC. Microscopically, these were associated with hemorrhage and/or presence of extracellular or intracellular (within macrophages) foreign material presumed to represent predominantly adjuvant/test article. The lesions were therefore considered consistent with an expected local reaction to foreign material at the injection sites. Upon recovery (4 weeks after injection), no macroscopic findings related to the administration of poly-ICLC were noted. Despite differences between the skin of non-human primates to human skin, we expect to find similar transient cellular infiltration at the site of poly ICLC s.c. injection.

In addition to its role in anti tumor and viral immunity mentioned above, topical imiquimod has been used as an adjuvant in combination with intradermal NY-ESO-1 protein in melanoma patients. This combination induced dermal mononuclear cell infiltrates in all patients. The infiltrates were composed primarily of T cells, monocytes, macrophages, myeloid DCs, NK cells, and, to a lesser extent, plasmacytoid DCs (Adams et al., 2008). Poly ICLC however acts on different PRRs, MDA-5 and TLR-3, and likely induces secretion of type-I IFNs locally. In situ immunomodulatory effects of poly ICLC are likely to differ from the effects of imiquimod. Combining immunohistochemistry evaluation of the cellular infiltrates induced by poly ICLC along with gene array analysis of its transcriptional effects on whole skin from the injection site may help elucidate the local events and mechanisms whereby poly ICLC exerts an adjuvant effect.

By working with our collaborator, Rafick Sekaly, who has used systems biology to monitor innate and adaptive responses to yellow fever vaccine and other patient cohorts (Gaucher et al., 2008), we can understand adjuvant perturbation of immune function. Blood and skin samples collected from the study volunteers will be sent to Dr. Sekaly's lab at the Vaccine and Gene Therapy Institute, where transcriptional arrays and high order bioinformatics analyses will be performed to obtain a global understanding of the innate immune responses to poly ICLC.

The proposed study is an open label study to evaluate the innate immune responses induced poly ICLC in healthy volunteers. The objectives of the study are to characterize the transcriptional changes induced by subcutaneous administration of poly ICLC on different blood cell types and to characterize the cellular infiltrates and transcriptional changes at the site of poly ICLC injection.

Primary Hypothesis Administration of poly ICLC to healthy volunteers will induce distinct transcriptional changes in different blood cell types, including different subsets of DCs.

Secondary Hypothesis Administration of poly ICLC to healthy volunteers will induce distinct transcriptional changes, and T cell and myeloid cell infiltrate in the skin at the site of injection.

Primary Aim:

To evaluate the innate immune responses to poly ICLC in different blood cell types, including three subsets of dendritic cells after subcutaneous administration to healthy volunteers.

Secondary Aims:

* To evaluate the innate immune responses to poly ICLC at the injection site.
* To evaluate the reproducibility of innate immune responses in whole PBMCs after a second dose of poly ICLC, in volunteers who participated in protocol MAC-682 and now return to participate in this proposed study.

Primary Outcome(s):

* Transcriptional arrays in whole PBMCs and in 8 subsets of blood leukocytes (naïve and memory T, NK, B, monocytes and three different subsets of dendritic cells (BDCA1+, BDCA3+ and BDCA2+ plasmacytoid DCs) following s.c. administration of poly ICLC.
* Flow cytometric analysis of activation markers in different subsets of blood leukocytes.
* Measurement of cytokines in the serum and/or plasma following s.c. administration of poly ICLC.

Secondary Outcome(s):

* Routine histology and immunohistochemistry to evaluate cellular infiltrates following subcutaneous injection of poly ICLC.
* Transcriptional analysis of skin samples from study drug injection site and from a non-lesional site of skin.
* Transcriptional analysis of whole PBMC samples at different timepoints following the first dose and the second dose of poly ICLC in volunteers who participated in protocol MAC-682 and are now returning to participate in this proposed study.

Methods and Procedures:

Pre-Screening Questionnaire Potential participants will first undergo pre-screening by telephone to assess medical history and qualification for the study (Appendix C - Pre-screening Questionnaire). Potential volunteers will have the opportunity to discuss the study and ask questions of the study recruiter at this time. Those who are eligible and interested in participation will attend a screening visit at the Rockefeller Hospital Outpatient Clinic.

Screening Visit

During the screening visit, study personnel will answer any questions about the study. Written informed consent will be obtained prior to conducting any study procedures. To ensure informed consent, the principal investigator or designee will discuss the following processes and explanations individually with each volunteer:

1. Pre HIV-test counseling.
2. Sexually active volunteers should use a reliable form of contraception from screening until 6 weeks after drug administration.

If the volunteer consents to participate, site personnel will:

* Perform complete medical history (including concomitant medication);
* Perform a general physical examination including height, weight, vital signs (pulse, respiratory rate, blood pressure and temperature), examination of skin, respiratory, cardiovascular and abdominal systems, and an assessment of cervical and axillary lymph nodes;
* Collect blood and urine specimens for all tests as indicated in the Schedule of Procedures (Appendix A);
* Perform a pregnancy test for all female volunteers.

Screening laboratory test(s) may be repeated at the discretion of the principal investigator or designee to investigate any isolated abnormalities.

If the screening visit occurs more than 45 days prior to date of drug administration, then study procedures for the screening visit must be repeated. However, the complete medical history may be replaced by an interim medical history and the informed consent form may be reviewed without signing again.

Drug Administration Visit (Day 0)

Prior to the study drug administration, site personnel will:

* Answer any questions about the study;
* Review interim medical history (including concomitant medications);
* Review safety laboratory data;
* Review the informed consent form administered at screening visit with volunteer;
* Perform a directed physical examination including vital signs (pulse, respiratory rate, blood pressure and temperature) as well as an assessment of axillary lymph nodes and any further examination indicated by history or observation;
* Collect blood and urine specimens for all tests as indicated in the Schedule of Procedures (Appendix A);
* Perform a pregnancy test for all female volunteers (blood will be sent stat) and obtain results prior to drug administration
* Perform baseline assessment of the site of study drug and evaluate and record any systemic symptoms;
* Administer study drug (sites of injection may be upper arms, thighs or buttocks)
* For volunteers who have agreed to undergo skin punch biopsies, two skin punch biopsies will be performed: one at a skin site contralateral to the injection site and the other at the injection site, 6 hours after study drug administration. The two selected skin sites for biopsy will be cleaned with povidone-iodine and anesthetized by injection of 1-2% of xylocaine. L.M.X.4 (Lidocaine 4%) a topical anesthetic cream may also be applied. Two punch biopsies of skin (6 mm) will be removed. The wounds will be sutured and sterile dressing applied. This procedure leaves a small and permanent scar.
* The volunteer will have the option to stay in the hospital overnight the night before study drug or placebo administration and/or the day of study drug administration for convenience ("boarders") or be scheduled as a day patient

Volunteers will be closely observed for at least 30 - 45 minutes after drug administration. Vital signs (pulse, respiratory rate, blood pressure and temperature) will be monitored at 30 - 45 minutes after vaccination and recorded. Any local and systemic reactogenicity events, as well as any other event that occurs, will be recorded at 30 - 45 minutes. Volunteers will be given a diary card (Appendix B) and asked to record any reactogenicity events that occur in first day after drug administration and between days 1 and 3 and between days 3 and 7. Site staff will explain to the volunteer how to record reactogenicity events.

Medical photography will be done to document the injection site and changes post injection, if any. The volunteer's identity will be kept confidential.

Day 1 Post-Drug Administration Visit

* Review of interim medical history and use of concomitant medications;
* If symptoms are present, perform a symptom-directed physical examination;
* Assess local and systemic reactogenicity as well as any other adverse events;
* Collect blood and urine specimens for all tests as indicated in the Schedule of Procedures (Appendix A).
* For volunteers who have agreed to undergo skin punch biopsies, one additional skin punch biopsy will be performed 1 day after study drug administration, at the injection site. The selected skin site for biopsy will be cleaned with povidone-iodine and anesthetized by injection of 1-2% of xylocaine. L.M.X.4 (Lidocaine 4%) a topical anesthetic cream may also be applied. One punch biopsy of skin (6 mm) will be removed. The wound will be sutured and sterile dressing applied. This procedure leaves a small and permanent scar.

Post-Drug Administration Visits

Volunteers will be asked to return to the clinic 2, 3, and 7 days after study drug administration. On those days the following will be conducted:

* Review of interim medical history and use of concomitant medications;
* If symptoms are present, perform a symptom-directed physical examination;
* Assess local and systemic reactogenicity as well as any other adverse events;
* Collect blood and urine specimens for all tests as indicated in the Schedule of Procedures (Appendix A);

Follow Up Visit

At Week 2, volunteers will be asked to return to the clinic for an additional assessment of safety and immunogenicity. The following will be conducted at this visit:

* Review of interim medical history and use of concomitant medications;
* If symptoms are present, perform a symptom-directed physical examination;
* Assess any adverse events;
* Collect blood and urine specimens for all tests as indicated in the Schedule of Procedures (Appendix A);
* Suture removal after optional skin biopsies, if biopsies are performed.

Samples will not be shipped to our collaborator, Dr. Rafick Sekaly until his IRB approval is accepted and reviewed by Rockefeller's IRB.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 years on the day of screening and no greater than 60 years at the time of drug/placebo administration
2. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study (screening plus 2 weeks)
3. In the opinion of the principal investigator or designee, has understood the information provided. Written informed consent needs to be given before any study-related procedures are performed
4. Willing to undergo HIV testing and counseling, and receive HIV test results
5. If a sexually active male, willing to use an effective measure of contraception(condoms, anatomical sterility) throughout the study period and will be advised not to get his partner pregnant for 6 weeks after study drug administration
6. Females of child-bearing potential must agree to use one of the following methods of contraception for 2 weeks prior to date of screening evaluation through 6 weeks after study drug administration:

   Be surgically sterile Be abstinent (or willing to be) Use oral contraceptives, or other form of hormonal birth control including hormonal vaginal rings or transdermal patches Use an intra-uterine device (IUD) Use (by ensuring her male partner(s)uses)barrier contraception (condom) with spermicide Any other equivalent (as judged by the investigative team) methods of contraception
7. Healthy adult males and females, as assessed by a medical history, physical exam, and laboratory tests

Exclusion Criteria:

1. Allergy to lidocaine
2. Confirmed HIV-1 or HIV-2 infection
3. Any clinically significant abnormality on history or examination including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids, immunosuppressive, anticancer, or other medications considered significant by the trial physician within the last 6 months
4. Any clinically significant acute or chronic medical conditions requiring care of a physician (e.g., diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that in the opinion of the investigator would preclude participation
5. Any laboratory value outside of reference range, with the exception of any non-clinically significant Grade I elevations of liver function tests (AST, ALT, direct/total bilirubin), electrolytes (Na, K, Cl, CO2), Glucose, CBC, as determined by the Principal Investigator or his designee as well as creatinine if the estimated glomerular filtration rate is > 60 mL/min/1.73 m2
6. Confirmed diagnosis of hepatitis B (surface antigen, HbsAg); hepatitis C (HCV antibodies) or active syphilis
7. If female, pregnant, planning a pregnancy during the trial period or lactating
8. Receipt of a live attenuated vaccine within 30 days or other vaccine within 14 days of poly ICLC administration
9. Receipt of blood transfusion or blood products 6 months prior to drug administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the innate immune responses to poly ICLC in different blood cell types, including three subsets of dendritic cells after subcutaneous administration to healthy volunteers. | 2 years
  The variables to be assessed include:
  * Transcriptional arrays in whole PBMCs and in 8 subsets of blood leukocytes (naïve and memory T, NK, B, monocytes and three different subsets of dendritic cells (BDCA1+, BDCA3+ and BDCA2+ plasmacytoid DCs) following s.c. administration of poly ICLC.
  * Flow cytometric analysis of activation markers in different subsets of blood leukocytes.
  * Measurement of cytokines in the serum and/or plasma following s.c. administration of poly ICLC.

SECONDARY OUTCOMES:
To evaluate the reproducibility of innate immune responses in whole PBMCs after a second dose of poly ICLC, in volunteers who participated in protocol MAC-682 and now return to participate in this proposed study. | 2 years
  The following variable will be assessed:
  - Transcriptional analysis of whole PBMC samples at different timepoints following the first dose and the second dose of poly ICLC in volunteers who participated in protocol MAC-682 and are now returning to participate in this proposed study.
To evaluate innate immune responses to poly ICLC at the injection site. | 2 years
  The following will be assessed:
  * Routine histology and immunohistochemistry to evaluate cellular infiltrates following subcutaneous injection of poly ICLC.
  * Transcriptional analysis of skin samples from study drug injection site and from a non-lesional site of skin.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States